CLINICAL TRIAL: NCT07083037
Title: Enhancing Preschool Children's Attention and Behaviour: Parent-Focused Program
Acronym: BRIDGE-McGill
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: University of Manitoba (Other); Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Tasmia Hai, Assistant Professor, McGill University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-06-073; 430-2024-00718 (Other Grant/Funding Number: SSHRC)
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Maternal Depression; Self-Regulation, Emotion; Child Mental Disorder; Child Development; Attention Problems; Behaviour Problems; Parental Stress
Keywords: maternal depression; child attention problems; child behaviour problems; parental stress
MeSH Terms: conditions — Emotional Regulation; Neurodevelopmental Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: The study will recruit a group of caregivers who meet the current criteria for elevated symptoms of psychological distress as measured by a score of 5 and indicate symptoms to "somewhat cause difficulties" above on the Patient Health Questionnaire 9-item, AND who have children with elevated levels of attention and/or behavior problems as measured by a CBCL ADHD subscale T-Score score of > 65 OR confirmation of attention/behavior problems through a clinical interview. Eligible female caregivers (mothers, grandmothers, aunts, guardians) will be recruited, and the recruitment will occur concurrently over 12 weeks, will incorporate intervention materials from Dialectical Behavior Therapy (DBT) and parent skills training (BRIDGE).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRIDGE arm (Experimental): The BRIDGE program is a manualized therapy program that provides participants with parenting and DBT skills through video training modules and in-group sessions. Participants in the BRIDGE arm will participate in 12 weeks of 20-60-minute DBT and parenting skills training that will be delivered asynchronously via video (participants will access these by logging onto a password-protected website). The BRIDGE condition also includes weekly synchronous 1-hour virtual group therapy sessions as well as DBT and parenting skills worksheets to complete between sessions.
  Interventions: Behavioral: Building Regulation in Dual Generations (BRIDGE; DBT + Parenting)
- Support As Usual (No Intervention): Control group participants in the SAU arm will receive a list of local mental health and parenting resources, curated by our research team. Participants can access any intervention or resource participants would like throughout the duration of the program.

INTERVENTIONS:
Behavioral: Building Regulation in Dual Generations (BRIDGE; DBT + Parenting) — The BRIDGE intervention includes 12 weeks of 20-60-minute DBT and parenting skills training videos, delivered asynchronously via an online website requiring a participant login. Video content was drawn from concepts outlined in the DBT Skills Training Manual 2nd Edition (Linehan, 2015). Parenting videos will provide mothers with parenting skills education based on best practices in evidence-based positive parenting interventions (e.g., Parent Management Training, Positive Parenting, Kazdin, 1997; Sanders et al., 2014). The BRIDGE condition also includes weekly synchronous 1-hour virtual group therapy sessions and worksheets to complete weekly (as an opportunity to practice skill use).
  Arms: BRIDGE arm

SUMMARY:
This study aims to evaluate the feasibility and efficacy of the Building Regulation in Dual Generations (BRIDGE) program for caregivers with significant mental health concerns and preschool and young children (3-7 years old) with elevated attention and/or behavior problems. The BRIDGE program focuses on supporting parental psychological distress and improving young children's self-regulation (SR), thereby reducing their attention and behavior problems (Bridgett et al., 2015; Brikell et al., 2015; Landstedt and Almquist, 2019). The long-term goal of this work is to improve family well-being and social-emotional development for young children by implementing an accessible and scalable dual-regulation program. We will achieve this through the following key objectives:

1. Assess the feasibility and accessibility of BRIDGE for preschool and young children (3-7 years old) with significant attention and behavior programs through questionnaires asking about attendance, satisfaction, and unmet needs.
2. Examine the efficacy of BRIDGE compared to control group at improving maternal mental health and child attention and behavioral difficulties in young children (primary outcomes). We will also examine parenting stress (secondary outcome).
3. Identify predictors of academic readiness skills in preschool and young children. We hypothesize that an increase in parental and child emotion-regulation skills and reduced attention, as well as behavioral problems, will lead to increased pre-academic skills in children.

DETAILED DESCRIPTION:
Early exposure to parent psychological distress and mental health challenges (e.g. elevated depression, anxiety, sleep problems and parenting stress) is as a crucial risk factor for the development of children's own difficulties through the intergenerational transmission of maternal mental health framework (Landstedt and Almquist, 2019). The Building Regulation in Dual Generations (BRIDGE) program was designed to improve maternal mental health challenges (e.g. depression, anxiety, trauma, stress) and promote positive parenting thereby improving child behavior and mental health. It brings together evidence-based programs, including Dialectical Behavior Therapy (DBT), behavior management, emotion socialization and mindfulness parenting strategies, and has made significant improvement in maternal depression, as well as the mental health of their children, with greater changes observed in mothers with higher psychological distress (Penner-Goeke et al., 2023).

This project addresses a gap in the current literature by focusing on parent-focused support for preschool and young children with attention and behavior problems. It aims to empower parents with tools and strategies to positively impact their children's behavior. The expected contribution includes understanding effective family-focused supports that address both parental and child challenges early on, promoting positive family well-being. This research has broader implications for clinicians, educators and policymakers by offering practical strategies to improve young children's' behaviors and manage parental mental health challenges, ultimately enhancing overall child well-being and aligning with broader goals in child development and early education. The results will be disseminated through academic publication, and directly communicated within our network of community agencies, programs, clinics and school-systems in both Quebec, Ontario and Manitoba.

The current study will conduct a non-randomized parallel assignment feasibility pilot design to evaluate the feasibility and potential efficacy of the BRIDGE program in addressing parents' mental health difficulties and children's attentional and behavioral problems. We aim to recruit sixty parent-child dyads (30 participants and 30 controls) to take part in the study. Participants in the intervention group will complete the 12-week online BRIDGE program, along with in-person assessments at three time points: pre-intervention (week 0-1;T1), post-intervention (week 12; T2), and follow-up (3 months; T3). The control group will complete the same in-person assessments without participating in the intervention.

Our primary aim is to examine the feasibility of BRIDGE on maternal mental health and their children's mental wellbeing, executive functioning, and social-emotional development. Our secondary aims are to evaluate the efficacy of BRIDGE therapy in improving parenting stress and decreasing harsh parenting tendencies. Supplementary aims of this study include observing differences or changes for both mothers and children, in sleep quality, mental wellbeing, relationships, as well as child academic readiness before and after the BRIDGE program.

ELIGIBILITY:
Inclusion Criteria:

BRIDGE Therapy Group:

Participants are deemed eligible for the BRIDGE therapy group if they meet the following criteria:

1. Above the age of 18.
2. Self-identify as a mother of a child between the age of 3-7 years old.
3. Currently living in Quebec, Ontario, or Manitoba
4. Fluency in English.
5. Mothers must have clinically significant symptoms of depression (mild to moderate on the Patient Health Questionnaire and indicate symptoms to "somewhat cause difficulties") currently affecting them. Participants also need to report symptoms of depression during pregnancy or shortly after birth.
6. Their child has attention and/or behavior problems (T-score > 65 on the Child Behavior Checklist (CBCL) ADHD subscales) or confirmed attention and/or behavior problems through clinical interview.

Control Group:

Participants are deemed eligible for the Control group if they meet the following criteria:

1. Above the age of 18
2. Self-identify as a mother of a child between the age of 3-7 years old
3. Currently living in Quebec, Ontario, or Manitoba
4. Fluency in English or bilingual
5. Mothers must NOT have clinically significant symptoms of depression (mild to moderate on the Patient Health Questionnaire)
6. Their child DOES NOT have attention and/or behavior problems (T-score > 65 on the Child Behavior Checklist (CBCL) ADHD subscales).

Exclusion Criteria:

BRIDGE Therapy Group:

Participants were excluded if they A) did not meet the inclusion criteria listed above or B) were unable to attend the weekly BRIDGE group therapy sessions.

Furthermore, eligible participants were invited to complete a semi-structured intake interview with principal investigator (PI) Dr. Tasmia Hai or a graduate student trainee under Dr. Hai's supervision, during which further questions about their mental health and child behavior were asked to ensure their eligibility. Based on the clinical suitability interview, participants may be excluded if they are deemed to be ineligible based on A) the mother's absence of clinically significant mental health symptoms, and/or B) the child's absence of attention and/or behavior problems. When relevant, participants may be identified to participate in the control group instead if eligibility is met.

Control Group:

Participants were excluded if they did not meet the inclusion criteria listed above. Furthermore, eligible participants were invited to complete a semi-structured intake interview with principal investigator (PI) Dr. Tasmia Hai, during which further questions about their mental health and child behavior were asked to ensure their eligibility. Based on the clinical suitability interview, participants may be excluded if they are deemed to be ineligible based on a) the mother's presence of clinically significant mental health symptoms, and/or B) the child's presence of attention and/or behavior problems. When relevant, participants may be identified to participate in the BRIDGE therapy group instead if eligibility is met.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who self-identify as a mother or female primary caregiver (e.g., grandmothers raising grandchildren, gender diverse caregivers who identify as mothers) will be eligible to participate. The terms "mother" or "maternal" will be used throughout reports to describe all participants.
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in child mental illness symptoms | The CBCL 1.5-5 and 6-18 will be assessed during eligibility screening (T0), pre-intervention (T1), within a month following the intervention (T2), and at 3-month follow-up (T3).
  Changes in child mental illness symptoms will be assessed using the Child Behavior Checklist (CBCL) for ages 1.5-5 and 6-18. The CBCL is a parent-report questionnaire that measures child functioning across internalizing and externalizing symptoms. The CBCL contains 100 items, with scores ranging from 0-200. Higher scores indicated greater symptom severity. We will be analyzing changes in children's A) Total problem behaviors B) ADHD problems subscale scores C) Internalizing behaviors D) Externalizing Behaviors
Changes in parent report measures of their children's executive function skills | Assessed at pre-intervention (T1) and within a month following the intervention (T2), and at 3-month follow-up (T3).
  Changes in children's executive functioning skills will be measured using the Behavior rating Inventory of Executive Function - Preschool Edition (BRIEF-P) or Behavior rating Inventory of Executive Function - Second Edition. The BRIEF-P is a 63-item parent-report measure and it assesses executive functioning in young children (ages 2-5) across five key areas: Inhibit, Shift, Emotional Control, Working Memory, and Plan/Organize, evaluating skills such as impulse control, emotional regulation, flexibility, and memory for tasks. The BRIEF-2 is a 63-item parent-report measure and is designed for older children (ages 5-18). It includes similar scales, as well as additional ones such as Initiate, Self-Monitor, and Organization of Materials, to capture more complex executive functions required in school and daily life. Both provide index scores and a Global Executive Composite that reflects overall executive functioning.
Changes in maternal mental health symptoms | The PHQ-9 will be assessed during eligibility screening (T0) , pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  Depressive symptoms will be measured using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item self-report questionnaire with possible scores ranging from 0 to 27, with higher scores indicating greater symptom severity.
Program Engagement | Attendance is measured weekly throughout the 12-week program and immediately after the intervention (T2).
  Program engagement will be assessed in a variety of ways. Clinicians will take attendance during therapy sessions. At post-intervention, the investigators will ask participants to report on their use of the videos and homework assignments throughout the intervention. Participants will also complete a program acceptability questionnaire at post-intervention, which was created by the investigators for this project. The program acceptability questionnaire asks participants to rate how important various program components were to them and includes several open-ended questions for participants to describe their experiences in the program.

SECONDARY OUTCOMES:
Changes in parenting stress | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  Parenting stress will be measured using the Parenting Stress Index-Short Form (PSI-SF). The PSI-SF is a self-report questionnaire that requires respondents to answer questions regarding their overall experience with parenting stress using a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Scores range from 36-180. Higher scores indicate higher levels of stress.
Changes in harsh parenting | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  Harsh parenting will be measured using the Overreactivity subscale of the Parenting Scale (PS). The Overreactivity subscale contains 10 items related to harsh parenting behaviors. Harsh parenting includes expressing inappropriate anger, irritability, or meanness towards one's child. Totals scores range from 10 to 70, with higher scores indicating higher levels of harsh parenting.

OTHER OUTCOMES:
Changes in maternal anger | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  Changes in anger will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anger subscale. The subscale contains 5-items with scores ranging from 5-25. Higher scores indicate more anger.
Changes in maternal sleep problems | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  The Patient-Reported Outcomes Measurement Information System-Sleep Disturbance Subscale Short Form will be used to measure change in sleep disturbances. The subscale contains 8 items. Total scores range from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Changes in anxiety symptoms | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  Anxiety symptoms will be measured using the Generalized Anxiety Disorder 7-Item Scale (GAD-7). The GAD-7 contains 7 items with possible scores ranging from 0 to 21. Higher scores represent higher levels of anxiety symptoms.
Changes in ADHD Symptoms in parents | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  The Adult ADHD Self Report Scale (ASRS) will be used to measure attention problems and hyperactive behaviours in parents. The ASRS is an 18-item questionnaire that screens for ADHD symptoms in adults, based on DSM criteria. It includes two parts: Part A (6 questions) screens for the most predictive symptoms, while Part B adds more detail. Respondents rate how often they experience symptoms like inattention, impulsivity, and restlessness.
Changes in children's cognitive and language skills | Assessed at pre-intervention (T1), within a month following the intervention (T2) and at 3-month followup (T3).
  Subtests from the Kaufman Assessment Battery for Children, Second Edition Normative Update (KABC-II NU) will be used. The KABC-II NU is an individually administered test that measures the cognitive abilities of children ages 3-18. It focuses on assessing problem-solving skills, memory, and reasoning, with minimal reliance on verbal instructions. The core areas evaluated include sequential and simultaneous processing, planning, learning, and knowledge.
Changes in pre-academic skills | Assessed at pre-intervention (T1), within a month following the intervention (T2) and at 3-month followup (T3).
  The Bracken School Readiness Assessment, 4th Edition (BRSA-4) will be used to measure changes in academic readiness in children. The BSRA-4 is an individually administered test for children in preschool through second grade. It assesses core school readiness concepts such as color identification, knowledge of letters, numbers/counting ability, size and comparison words, and shape recognition. The BSRA-4 is developmentally sensitive and can help identify children who may need additional support before starting primary school. Scores reflect a child's exposure to basic academic concepts important for early learning.
Changes in parenting behaviors and practices | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  The Parenting Young Children Questionnaire (PARYC) will be used. The PARYC is a 21-item parent-report measure designed to assess parenting behaviors in parents of young children. It focuses on key domains such as setting expectations for behavior, supporting positive behavior, and managing misbehavior. Parents rate how often they use various effective parenting practices, which helps to identify strengths as well as areas where additional support or intervention may be needed.
Changes in maternal perceived social support | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  The Multidimensional Scale of Perceived Social Support (MSPSS) will be used to measure participant's levels of social support from significant others, family, and friends. Scores can range from 12-84. Higher scores indicated higher levels of perceived social support.
Changes in alcohol use | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  The Alcohol Use Disorder Identification Test (AUDIT) will be used to measure participants' use of alcohol. The AUDIT contains 10 questions and scores may range from 10 to 40. Higher scores indicate greater hazardous or harmful alcohol consumption.
Changes in cannabis use | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  The Cannabis Use Disorder Identification Test (CUDIT) will be used to measure participants' cannabis use. The scale contains 8 items. Scores may range from 0 to 32. Higher scores indicate more hazardous cannabis use.
Changes in recent stressful events (RSE) | Assessed at pre-intervention (T1), immediately after intervention (T2) and at 3-month follow-up (T3).
  The Recent Stressful Experiences checklist (RSE) was developed by study authors, based on recommendations from the JBP Research Network on Toxic Stress at the Harvard's Center on the Developing Child, to measure familial exposure to various stressors which may affect participants (2022). The scale contains two items which ask about various stressors that participants may have experienced. Each of these items' scores can range from 0 to 10, with higher scores indicating more stressful experiences. The scale also contains five items assessing participants' ability to cope with stressful events. Scores for these five questions range from 4-21, with higher scores indicating a greater ability to cope with stress.
Changes in difficulties with Emotion regulation | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  The Difficulties in Emotion Regulation Scale (DERS) will be used. The DERS is a 36-item self-report questionnaire that assesses problems with emotion regulation across six areas: nonacceptance of emotions, difficulty with goal-directed behavior, impulse control, lack of emotional awareness, limited access to regulation strategies, and lack of emotional clarity. Respondents rate how often each statement applies to them on a five-point scale, with higher scores indicating greater difficulties. The DERS is widely used to identify emotion regulation challenges and monitor changes over time in both clinical and research settings.
Changes in Children's Sleep Habits | Assessed at pre-intervention (T1), immediately after the intervention (T2), and at 3-month follow-up (T3).
  The Children's Sleep Habits Questionnaire will be used. The CSHQ is a 45-item parent-report tool that assesses common sleep problems in children aged 4-12 across eight areas, including bedtime resistance and night wakings. Items are rated based on frequency over the past week. Higher total scores indicate more severe sleep difficulties, with scores above 41 suggesting potential clinical concerns.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Manitoba - Department of Psychology, Winnipeg, Manitoba
  - McGill University - Department of Education and Counselling Psychology, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Proceedings of the 8th meeting of the European Pineal Society. Tours, France, 3-7 July 1999. Reprod Nutr Dev. 1999 May-Jun;39(3):275-408. No abstract available. PMID 10507827
- [Background] Leung CK, Shiu RP. Morphological and proliferative characteristics of human breast tumor cells cultured on plastic and in collagen matrix. In Vitro. 1982 May;18(5):476-82. doi: 10.1007/BF02796476. PMID 6749655
- [Background] Brikell I, Kuja-Halkola R, Larsson H. Heritability of attention-deficit hyperactivity disorder in adults. Am J Med Genet B Neuropsychiatr Genet. 2015 Sep;168(6):406-413. doi: 10.1002/ajmg.b.32335. Epub 2015 Jun 30. PMID 26129777
- [Background] Gwee AL. Brain drain. Med J Aust. 1974 Aug 17;2(2):suppl:20-1. No abstract available. PMID 4422221